CLINICAL TRIAL: NCT00495508
Title: A Randomised, Open-label Non-inferiority Trial of Artemether-lumefantrine Versus Quinine for the Treatment of Uncomplicated Falciparum Malaria During Pregnancy, Mbarara, Uganda (2006-2007)
Brief Title: Quinine vs. Artemether/Lumefantrine in Uncomplicated Malaria During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); University of Cape Town (Other); Shoklo Malaria Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mba/06/MIP
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2019-08

CONDITIONS: Malaria
Keywords: Quinine; Artemether; Lumefantrine; malaria; Uganda; Artemisinin- based combination therapy; pregnancy; Malaria In Pregnancy
MeSH Terms: conditions — Malaria | interventions — Quinine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quinine (Active Comparator)
  Interventions: Drug: Quinine
- Arthemeter lumefantrine (Active Comparator)
  Interventions: Drug: artemether / lumefantrine

INTERVENTIONS:
Drug: Quinine
  Arms: Quinine
Drug: artemether / lumefantrine
  Arms: Arthemeter lumefantrine

SUMMARY:
A) for the treatment of uncomplicated malaria during second and third trimester pregnancy to oral Quinine hydrochloride. The PCR-corrected adequate clinical and parasitological response (ACPR) on day 42 is considered as the primary efficacy criterion. Newborns will be followed for growth and development indicators.

DETAILED DESCRIPTION:
Study Title:

Efficacy and Safety of Quinine vs Artemether/Lumefantrine in uncomplicated malaria during pregnancy, Mbarara, Uganda (2006/2007).

Regulatory Status:

Investigational - Phase IV

Investigational Product and route:

* Quinine hydrochloride, oral route.
* Coartem® (Novartis Pharma AG, Basel, Switzerland), oral route.

Lead Investigator and Study Centre Primary objective - To establish that, in pregnant women with uncomplicated Plasmodium falciparum malaria, the PCR-adjusted efficacy of Artemether/Lumefantrine is not inferior to oral Quinine.

Secondary objectives

* To define the pharmacokinetics of the combination artemether-lumefantrine (AL) in the treatment of uncomplicated P. falciparum infections in the last two trimesters of pregnancy.
* To collect baseline data on maternal, obstetric and infant outcomes.
* To estimate the incidence of malaria infection, both microscopic and sub-microscopic (by PCR) during pregnancy.
* women attending Mbarara National Referral Hospital (MNRH) ante-natal clinic (ANC).
* Women with a positive blood smear during follow-up will be invited to participate in a non-inferiority, open, randomised, non- inferiority trial comparing the efficacy and tolerance of Coartem® (Artemether-Lumefantrine) for the treatment of uncomplicated malaria during second and third trimester pregnancy to oral Quinine hydrochloride. PCR-corrected adequate clinical and parasitological response (ACPR) on day 42 is considered as the primary efficacy criterion.
* Women with uncomplicated malaria from the efficacy study, will be followed to obtain an efficacy endpoint at 42 days OR at delivery, whichever timepoint is the last.
* Newborns will be followed monthly up to the age of 1 year.

Inclusion Criteria (Efficacy Study):

* Pregnant woman
* Malaria infection, detected by microscopy, with P. falciparum (mixed or mono-infection)
* Age of gestation: 13 weeks and beyond
* Efficacy study signed informed consent form

Exclusion Criteria (Efficacy Study):

* P. falciparum parasitaemia above 250,000 parasites/μl
* Severe anaemia
* Signs or symptoms of severe/complicated malaria requiring parenteral treatment (WHO 2000)
* Known allergy to artemisinin derivatives, lumefantrine or quinine;
* Previous participation in the efficacy study
* Inability to attend the efficacy study follow-up schedule.

Study drugs and Administration

* Group 1 (Active Control): Quinine hydrochloride (10 mg/Kg/8h for 7 days) administered orally.
* Group 2 (Test): Coartem®, fixed Artemether-Lumefantrine (20/120 mg) GMP manufactured by Novartis Pharma AG (Basel, Switzerland), 4 tablets twice a day for 3 days with 200 ml of milk tea at each dose .

Endpoints

- Primary efficacy endpoint: PCR-corrected adequate clinical and parasitological response (ACPR) on Day 42.

* Secondary efficacy endpoints:
* PCR-corrected(ACPR)at delivery
* Pharmacokinetic parameters
* Symptom clearance Time
* Proportion of patients who have fever cleared at Day 1, 2 and 3
* Safety endpoints:
* Incidence of any adverse events
* Pregnancy outcome
* Infant development during the first year of life

ELIGIBILITY:
Inclusion Criteria:

Cohort Study:

* Weeks of pregnancy between 13 and 22 weeks
* Resident in Mbarara Municipality (radius of 15km from MNRH)
* Cohort study signed informed consent form

Efficacy Study:

* Pregnant woman
* Malaria infection, detected by microscopy, with P. falciparum (mixed or mono-infection)
* Age of gestation: 13 weeks and beyond
* Efficacy study signed informed consent form

Exclusion Criteria:

Efficacy Study:

* P. falciparum parasitaemia above 250,000 parasites/μl
* Severe anaemia
* Signs or symptoms of severe/complicated malaria requiring parenteral treatment (WHO 2000)
* Known allergy to artemisinin derivatives, lumefantrine or quinine;
* Previous participation in the efficacy study
* Inability to attend the efficacy study follow-up schedule.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PCR-corrected adequate clinical and parasitological response (ACPR) on Day 42 or at delivery. | 3 years

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 3.5 years
Incidence of adverse events | 3 years
Pregnancy outcome | 3.5 years
Infant development during the first year of life | 3 years
Histopathological findings in the placenta | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Piola, MD, MPH, Principal Investigator — Epicentre; Philippe J Guerin, MD, MPH, PhD, Study Chair — Epicentre; Elizabeth Ashley, MB BS, Study Chair — Epicentre; Rose McGready, MD, PhD, Study Chair — Shoklo Malaria Research Unit (SMRU); François Nosten, MD, PhD, Study Chair — SMRU
Locations (1):
- Epicentre, Mbarara, Mbarara District, Uganda

REFERENCES:
- [Derived] De Beaudrap P, Turyakira E, Nabasumba C, Tumwebaze B, Piola P, Boum Ii Y, McGready R. Timing of malaria in pregnancy and impact on infant growth and morbidity: a cohort study in Uganda. Malar J. 2016 Feb 16;15:92. doi: 10.1186/s12936-016-1135-7. PMID 26879849
- [Derived] De Beaudrap P, Turyakira E, White LJ, Nabasumba C, Tumwebaze B, Muehlenbachs A, Guerin PJ, Boum Y, McGready R, Piola P. Impact of malaria during pregnancy on pregnancy outcomes in a Ugandan prospective cohort with intensive malaria screening and prompt treatment. Malar J. 2013 Apr 24;12:139. doi: 10.1186/1475-2875-12-139. PMID 23617626
- [Derived] Muehlenbachs A, Nabasumba C, McGready R, Turyakira E, Tumwebaze B, Dhorda M, Nyehangane D, Nalusaji A, Nosten F, Guerin PJ, Piola P. Artemether-lumefantrine to treat malaria in pregnancy is associated with reduced placental haemozoin deposition compared to quinine in a randomized controlled trial. Malar J. 2012 May 3;11:150. doi: 10.1186/1475-2875-11-150. PMID 22554092
- [Derived] Piola P, Nabasumba C, Turyakira E, Dhorda M, Lindegardh N, Nyehangane D, Snounou G, Ashley EA, McGready R, Nosten F, Guerin PJ. Efficacy and safety of artemether-lumefantrine compared with quinine in pregnant women with uncomplicated Plasmodium falciparum malaria: an open-label, randomised, non-inferiority trial. Lancet Infect Dis. 2010 Nov;10(11):762-9. doi: 10.1016/S1473-3099(10)70202-4. PMID 20932805